CLINICAL TRIAL: NCT03649464
Title: A Phase Ib/2 Open-label Study Investigating the Tolerability, Safety, Pharmacokinetic Properties and Efficacy of Oral OKN-007 in Participants With Recurrent High-grade Glioma
Brief Title: Investigation of Oral OKN-007 in Recurrent High-grade Glioma Participants
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Planned to execute the new Oral OKN-007 clinical trial with modified study plan soon. This Study not proceeding and sites never opened.
Sponsor: Oblato, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OKN-007-OL-RMG-201
Record Dates: First submitted 2018-08-17; First posted 2018-08-28 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma; Astrocytoma; Oligodendroglioma
Keywords: recurrent high-grade glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma | interventions — OKN 007

STUDY DESIGN:
Intervention Model Description: Dose escalation cohort: 1000mg twice daily (BID), 1000mg thrice daily (TID), 1500mg thrice daily (TID).
  Expansion cohort: MTD defined in the dose escalation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OKN-007 (Experimental): Oral OKN-007
  Interventions: Drug: OKN-007

INTERVENTIONS:
Drug: OKN-007 — Dose escalation/PK cohort (Phase Ib): 1000mg twice daily (BID), 1000mg thrice daily (TID), 1500mg thrice daily (TID).
  Expansion cohort (Phase 2): MTD defined in the dose escalation (Phase Ib) study.
  Other Names: Anti-Cancer Agent

SUMMARY:
The objective of this study is to investigate tolerability, safety, pharmacokinetics (PK) and efficacy of oral OKN-007 in participants with recurrent high-grade glioma.

DETAILED DESCRIPTION:
Dose escalation/PK study (Phase Ib) will follow a traditional 3+3 design with evaluable participants enrolled at each dose level: Cohort 1 (1000mg, BID), Cohort 2, (1000mg, TID), and Cohort 3 (1500 mg, TID). The food-effect study will be one-week add-on study at the beginning of the dose escalation/PK study. Dose expansion study (Phase 2) will proceed to treat at the maximum tolerated dose (MTD) up to 2 years or until tumor progression, unacceptable toxicity, death or participants withdrawal. Participant may continue receiving treatment beyond 2 years at the discretion of investigator.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathology of recurrent gliomas that were originally diagnosed as, Glioblastoma (WHO Grade IV), Astrocytoma (WHO Grade III), or Oligodendroglioma (WHO Grade III). Participants with an initial diagnosis of a lower-grade glioma are eligible if a subsequent biopsy was determined to be glioblastoma.
* Unequivocal radiographic evidence of tumor progression by MRI as per the RANO criteria within 14 days prior to registration.
* At least one measureable lesion per RANO.
* Prior radiotherapy
* Prior Temozolomide treatment, unless contraindications or intolerance.
* Last cytotoxic chemotherapy or biologic therapy treatment 14 or more days before study start (greater than or equal to 42 days if nitrosourea was administered).
* ECOG performance status of 0, 1 or 2.
* Full recovery (≤ grade 1) from the toxic effects of any earlier intervention and a minimum of 28 days from the last administration of any investigational agent.
* Adequate renal, liver and bone marrow function: Leukocytes >3,000/mcL; Absolute neutrophil count >1,500/mcL; Platelets >100,000/mcL; Total bilirubin ≤ 1.5 x ULN; AST (SGOT) / ALT (SGPT) ≤ 2.5 x ULN; Creatinine clearance ≥ 60 mL/min calculated as per Cockcroft-Gault equation.
* Must be ≥ 18 years of age.
* Life expectancy (as assessed by the Investigator) at least three months.
* Capability of swallowing oral medication (4-6 size 0 capsules twice or thrice a day).
* Have provided verbal and written informed consent.
* Must be willing to have multiple blood draws for PK analysis.
* Female participants, of childbearing potential, must have a negative serum pregnancy test within 72 hours of taking study medication and agrees to abstain from activities that could result in pregnancy from enrollment through 120 days after the last dose of study treatment.
* Male participants must agree to use an adequate method of contraception.

Exclusion Criteria:

* Second primary malignancy expected to require treatment within a 6 month period (except adequately treated basal cell carcinoma of the skin). Participants who had another malignancy in the past, but have been free of active disease for more than 2 years, are eligible.
* Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the Investigator, would compromise the safety of the participants and his/her ability to complete the study.
* with abnormal sodium, potassium, or creatinine levels ≥ grade 2.
* with PT/PTT or INR above the upper limit of normal, unless treated with anticoagulants (e.g. warfarin). In such cases coagulation parameters (INR) should be monitored weekly for the first six weeks of the study.
* Inability to comply with protocol or study procedures.
* Women who are pregnant or breastfeeding.
* For participation in a food effect cohort, uncontrolled Diabetes Type I or uncontrolled Type II (HbA1c > 7 mmol/L assessed locally) as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with DLTs (Dose Limiting Toxicities) and AEs (Adverse Events) | 28 days
  It will be summarized by dose cohort and by overall safety evaluable population using CTCAE v5.0 for Phase Ib dose escalation and Phase 2 dose expansion cohort.
Number of Participants with Best Overall Response Rate in the brain | 24 months
  The rate of participants with complete response of partial response using Response Assessment in Neuro-Oncology Criteria (RANO) will be summarized for Phase 2 dose expansion cohort.

SECONDARY OUTCOMES:
Proportion of Participants as Assessed by 6-month Progression-Free Survival (PFS) | 6 months
  Proportion of participants who are progression free after six months will be calculated for Phase Ib dose escalation and Phase 2 dose expansion cohort.
Proportion of Participants as Assessed by Overall Survival (OS) | 24 months
  Proportion of participants who are alive will be calculated as the time (days) from Day 1 to the participant's death for Phase Ib dose escalation and Phase 2 dose expansion cohort.
The Cmax of OKN-007 in plasma | Day 1 and Day 14
  Blood samples will be collected at 10 time points during the 47.5 hours for Phase Ib dose escalation cohort.
The Tmax (time to maximum concentration) of OKN-007 in plasma | Day 1 and Day 14
  Blood samples will be collected at 10 time points during the 47.5 hours for Phase Ib dose escalation cohort.
AUC (area under the time curve) of OKN-007 in plasma | Day 1 and Day 14
  Blood samples will be collected at 10 time points during the 47.5 hours for Phase Ib dose escalation cohort.
Plasma concentration of OKN-007 | Before the first dose on Day 8 and before the first dose of Day 29 in the morning
  Blood samples will be collected for participants enrolled in Phase 2 expansion cohort.
OKN-007 plasma levels over time for food-effect study | Day 7 and Day 4 before the beginning of the dose escalation/PK study
  Blood samples will be collected on prior to dosing and at the following samples after OKN-007 single dose during 47.5 hours for participants enrolled in the food-effect study in Phase Ib dose escalation cohort.

IPD SHARING:
Plan to Share IPD: No